CLINICAL TRIAL: NCT00950729
Title: The Effects of Lower Right Limb Orthopedic Immobilization on Driving Performance: an Experimental Study During Simulated Driving in Healthy Volunteers.
Brief Title: The Effects of Lower Right Limb Orthopedic Immobilization on Driving Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: BSN Medical Inc (Industry)
Responsible Party: Francois Cabana, Centre hospitalier universitaire de Sherbrooke (CHUS)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Socrate
Record Dates: First submitted 2009-03-02; First posted 2009-08-03 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Walking Cast Right Leg Immobilisation Effects; Aircast Right Leg Immobilisation Effects
Keywords: car driving simulator; orthopedic leg immobilisation; braking time; braking force
MeSH Terms: interventions — Casts, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Driving with Running Shoes (Active Comparator)
  Interventions: Procedure: Driving with running shoes
- Driving with Plaster cast (Active Comparator)
  Interventions: Procedure: Plaster cast
- Driving with Aircast (Active Comparator)
  Interventions: Procedure: Driving with Aircast

INTERVENTIONS:
Procedure: Driving with running shoes — Participant was asked to do all the experiments with their own running shoes
  Arms: Driving with Running Shoes
Procedure: Plaster cast — The participant was ask to do all the experiments with a plaster cast molded on his right leg
  Arms: Driving with Plaster cast
Procedure: Driving with Aircast — The participant was ask to do all the experiments with a aircast on his right leg
  Arms: Driving with Aircast

SUMMARY:
Abstract Background: Effects of orthopedic immobilizations of the lower right limb on driving performances are unknown. Therefore, clinicians and legislators cannot put forth recommendations for road safety for patients requiring such immobilizations. The objective of the present study was to evaluate the effects of different orthopedic immobilizations on braking performances in simulated driving conditions.

Methods: The braking performances of 48 healthy volunteers were evaluated under 3 conditions: wearing their running shoes, and 2 types of orthopedic immobilizations of the lower right limb, a walking cast and an Aircast walker. A computerized driving simulator was used to measure the maximum force applied on the brake pedal during braking, the braking reaction time and the total braking time during emergency braking with and without a distracter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 25 and 60 years old
* Valid Québec driving license
* Driving for at least five years
* Must used exclusively the right foot for accelerating and braking

Exclusion Criteria:

* Non-compensated visual acuity deficits or other visual problems
* Drug or alcohol abuse
* Use of psychotropic drugs
* Central nervous system illnesses such as epilepsy
* Sleep issues
* Metabolic problems
* Cardiovascular disease
* Cerebrovascular disease
* Peripheral vascular disease
* Psychiatric illness
* Renal disease
* Musculoskeletal disease
* Motion sickness and
* Simulator sickness

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: François Cabana, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Research Centre on Aging, Sherbrooke Geriatric University Institute (IUGS),, Sherbrooke, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: march 2007 to june 2007 recruitment was done at the CHUS
Period: Driving With Running Shoes
Arm/Group | Healthy Subjects
Started | 48 (March 2007)
Completed | 48 (June 2007)
Not Completed | 0
Period: Driving With Plaster Cast
Arm/Group | Healthy Subjects
Started | 48
Completed | 48
Not Completed | 0
Period: Driving With Aircast
Arm/Group | Healthy Subjects
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.27 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 24
Region of Enrollment [Number; unit: participants]
  Canada | 48

OUTCOME MEASURES:

1. Primary Outcome: Mean Breaking Time Measured on a Driving Car Simulator
Description: computerized driving simulator was used to measure the braking reaction time and the total braking time during emergency braking with and without a distracter.
Time Frame: June 2007 to September 2007
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 48
seconds | 0.58 (.041)

2. Primary Outcome: Mean Breaking Force Measured on a Driving Car Simulator
Description: computerized driving simulator was used to measure the braking force during emergency braking with and without distractor
Time Frame: June 2007 to September 2007
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 48
pounds | 293.8 (75.2)

ADVERSE EVENTS:
Arm/Group | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes